CLINICAL TRIAL: NCT04260919
Title: Chest Physiotherapy in Light and Moderate Bronchiolitis in Ambulatory Children Under Two Years of Age - a Randomised Control Trial
Brief Title: Chest Physiotherapy in Bronchiolitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Responsible Party: Principal Investigator, Frederico Ramos Pinto, Principal Investigator, Universidade do Porto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FRP-01
Record Dates: First submitted 2020-02-06; First posted 2020-02-07 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Bronchiolitis
Keywords: bronchiolitis; chest physiotherapy; children
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Intervention Model Description: Randomized trial with two groups.
Masking Description: One control group and one intervention group, where chest physiotherapy is used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The participants just received standard medical treatment
- Intervention (Experimental): The participants received medical treatment and chest physiotherapy sessions
  Interventions: Procedure: Chest physiotherapy

INTERVENTIONS:
Procedure: Chest physiotherapy
  Arms: Intervention

SUMMARY:
Randomized trial of chest physiotherapy in outpatients with bronchiolitis under two years of age, during two consecutive seasonal outbreaks.

DETAILED DESCRIPTION:
A randomized controlled trial was conducted (following CONSORT Statement) in the Paediatric Emergency Department of Centro Hospitalar Universitário São João-Porto (CHUSJ), a tertiary care hospital, during the period from December to March in 2011 and 2012.

Ethical approval was obtained from the Ethics Committee of Centro Hospitalar Universitário São João-Porto.

Children up to 2 years of age, both genders, with a diagnosis of acute bronchiolitis based on clinical findings, including wheezing or wheezing with crackles, respiratory distress and alteration of feeding condition, were signalized by the physician who met them at the emergency room.

Then, the main investigator of the study interviewed the caregivers and informed about the aims and procedures of the study, after a formal written consent in accordance with the Declaration of Helsinki was sign by all the caregivers.

Severity grade was established with the Kristjansson Respiratory Score which variate from light to severe, being the light to moderate selected to study.

Randomization in intervention or control group was made by the method of permuted-blocks. All children were assessed in a calm environment, while awake and not crying, and were submitted to a standard assessment protocol consisting of a clinical demographic data collection by interview of parents and the application of the Kristjansson Respiratory Score. All children underwent the same medical treatment protocol at the pediatric emergency department (PED), consisting in nebulization with medication, during the emergency room episode, and counselled in the subsequent one or two weeks and were followed during two weeks after discharge from PED, being reassessed at the end of the two weeks.

Children from Intervention Group (IG) underwent a standard intervention chest physiotherapy protocol performed by a physiotherapist, consisting on the techniques: prolonged slow expiration (PSE), rhinopharyngeal retrograde clearance (RRC) and provoked cough (PC).

ELIGIBILITY:
Inclusion Criteria:

* Children up to 2 years of age, both genders, with a diagnosis of acute bronchiolitis

Exclusion Criteria:

* presence of comorbidities, such as cystic fibrosis, neuromuscular, congenital heart disease, prematurity or respiratory distress and all the cases that were admitted into the hospital

Ages: 15 Days to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2011-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Reduction of Kristjansson Respiratory Score | Baseline; after two weeks of treatment
  Verified by changes in the Kristjansson Respiratory Score, which is a practical and simple score, that assesses the main signs and symptoms of bronchiolitis, having a good validity and inter-observer reliability.It assigns a value between 0 and 2 to each of the five variables: respiratory rate, chest recession, breath sound, skin colour and general condition. A higher Kristjansson respiratory score indicate a worse respiratory condition.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roque-Figuls M, Gine-Garriga M, Granados Rugeles C, Perrotta C, Vilaro J. Chest physiotherapy for acute bronchiolitis in paediatric patients between 0 and 24 months old. Cochrane Database Syst Rev. 2023 Apr 3;4(4):CD004873. doi: 10.1002/14651858.CD004873.pub6. PMID 37010196
- [Derived] Pinto FR, Alexandrino AS, Correia-Costa L, Azevedo I. Ambulatory chest physiotherapy in mild-to-moderate acute bronchiolitis in children under two years of age - A randomized control trial. Hong Kong Physiother J. 2021 Dec;41(2):99-108. doi: 10.1142/S1013702521500098. Epub 2021 Mar 31. PMID 34177198
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3433974/
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/23287014